CLINICAL TRIAL: NCT00721253
Title: Visual Outcomes of Subjects Bilaterally Implanted With ReSTOR Aspheric +4 vs. Tecnis Multifocal Intraocular Lens (IOL) or Acri.LISA IOL
Brief Title: Visual Outcomes of Subjects Bilaterally Implanted With ReSTOR Aspheric +4 vs. Tecnis or Acri.LISA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Rick Potvin, Alcon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M07-002
Record Dates: First submitted 2008-07-21; First posted 2008-07-24 (Estimated); Results first posted 2010-03-16 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Cataract
Keywords: ReSTOR
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- ReSTOR Aspheric +4 (Active Comparator): ACRYSOF ReSTOR Aspheric +4 Model SN6AD3
  Interventions: Device: ReSTOR
- Tecnis MF (Active Comparator): Abbott Medical Optics Tecnis Multifocal Intraocular Lens (IOL) Model ZM900
  Interventions: Device: Tecnis
- Acri.LISA (Active Comparator): Meditec Acri.LISA Intraocular Lens (IOL) Model 366D
  Interventions: Device: Acri.LISA

INTERVENTIONS:
Device: ReSTOR — Implantation of the ReSTOR Aspheric +4 (SN6AD3) multifocal intraocular lens (IOL)
  Arms: ReSTOR Aspheric +4
Device: Tecnis — Implantation with the Tecnis multifocal (ZM900) intraocular lens (IOL)
  Arms: Tecnis MF
Device: Acri.LISA — Implantation with the Acri.LISA 366D multifocal intraocular lens (IOL)
  Arms: Acri.LISA

SUMMARY:
This is a study to compare visual outcomes of subjects bilaterally implanted w/ReSTOR to subjects bilaterally implanted with the Tecnis Multifocal Intraocular Lens (IOL) or Acri.LISA IOL

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cataracts

Exclusion Criteria:

* Preexisting condition likely to confound results; 1 D astigmatism by preoperative K-readings

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects 18 years or older of either sex and any race; bilateral diagnosis of cataracts.
  There were no patients that received implantation of the Tecnis Multifocal lens.
Pre-assignment Details: Subject eligibility was determined at the pre-operative visit.
Groups:
- ReSTOR Aspheric +4: Bilateral implantation of ACRYSOF ReSTOR Aspheric +4 Model SN6AD3
- Acri LISA IOL: Bilateral Implantation of Meditec Acri.LISA Intraocular Lens (IOL) Model 366D
Period: Overall Study
Arm/Group | ReSTOR Aspheric +4 | Acri LISA IOL | Tecnis MF
Started | 20 | 22 | 0 (There were no subjects that were implanted with the Tecnis lens.)
Completed | 20 | 22 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ReSTOR Aspheric +4 | Acri LISA IOL | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 21 | 33
  >=65 years | 8 | 1 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Uncorrected Visual Acuity (UCVA) at Distance, Near and Intermediate
Description: Uncorrected Visual Acuity (UCVA) at distance, near and intermediate, measured in logMAR. LogMAR is the "logarithm of the minimum angle of resolution". It is a unit of measure for visual acuity (VA). A lower logMAR value indicates better visual acuity.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR Aspheric +4 | Acri LISA IOL
Number analyzed (Participants) | 20 | 22
logMAR
  UCVA 4 m | 0.02 (0.13) | 0.01 (0.18)
  UCVA 80 cm | 0.20 (0.14) | 0.20 (0.15)
  UCVA 60 cm | 0.21 (0.14) | 0.19 (0.14)
  UCVA Near at 40 cm | -0.04 (0.18) | -0.05 (0.07)

2. Secondary Outcome: Contrast Sensitivity
Description: Contrast sensitivity is the measurement of one's ability to detect slight changes in luminance before it becomes indistinguishable. It is measured in logarithmic units by means of an illuminated box, the CSV 1000 by Vector Vision. A higher value for the logarithmic units translates to better contrast sensitivity.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: log units
Arm/Group | ReSTOR Aspheric +4 | Acri LISA IOL
Number analyzed (Participants) | 20 | 22
log units
  Contrast Sensitivity 1.5 cpd (cycles per degree) | 1.88 (0.20) | 1.78 (0.27)
  Contrast Sensitivity 3 cpd | 1.98 (0.23) | 2.01 (0.15)
  Contrast Sensitivity 6 cpd | 1.94 (0.24) | 1.99 (0.16)
  Contrast Sensitivity 12 cpd | 1.57 (0.31) | 1.53 (0.22)
  Contrast Sensitivity 18 cpd | 1.02 (0.42) | 1.07 (0.30)
  Mesopic Conditions, 1.5 cpd | 1.87 (0.21) | 1.83 (0.15)
  Mesopic Conditions, 3 cpd | 1.91 (0.22) | 1.83 (0.16)
  Mesopic Conditions, 6 cpd | 1.68 (0.23) | 1.62 (0.25)
  Mesopic Conditions, 12 cpd | 1.11 (0.36) | 1.16 (0.36)
  Mesopic Conditions, 18 cpd | 0.54 (0.26) | 0.52 (0.22)
  Mesopic Conditions w/glare, 1.5 cpd | 1.56 (0.37) | 1.55 (0.31)
  Mesopic Conditions w/glare, 3 cpd | 1.56 (0.39) | 1.52 (0.24)
  Mesopic Conditions w/glare, 6 cpd | 1.31 (0.34) | 1.26 (0.24)
  Mesopic Conditions w/glare, 12 cpd | 0.72 (0.26) | 0.73 (0.19)
  Mesopic Conditions w/glare, 18 cpd | 0.34 (0.13) | 0.30 (0.00)

3. Secondary Outcome: Defocus Curve
Description: Defocus cureve. A defocus curve is created by multiple measurements of one's visual acuity at different spherical powers. Visual Acuity (VA) is measured in logMAR. LogMAR is the "logarithm of the minimum angle of resolution". A lower logMAR value indicates better visual acuity.
Time Frame: 6 months post-operative
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR Aspheric +4 | Acri LISA IOL
Number analyzed (Participants) | 20 | 22
logMAR
  Negative Defocus Curve, -5.0 Diopter | 0.55 (0.13) | 0.58 (0.12)
  Negative Defocus Curve, -4.5 Diopter | 0.38 (0.10) | 0.42 (0.13)
  Negative Defocus Curve, -4.0 Diopter | 0.24 (0.14) | 0.27 (0.12)
  Negative Defocus Curve, -3.5 Diopter | 0.08 (0.08) | 0.08 (0.11)
  Negative Defocus Curve, -3.0 Diopter | 0.0 (0.08) | 0.02 (0.09)
  Negative Defocus Curve, -2.5 Diopter | 0.09 (0.12) | 0.08 (0.11)
  Negative Defocus Curve, -2.0 Diopter | 0.29 (0.13) | 0.27 (0.16)
  Negative Defocus Curve, -1.5 Diopter | 0.31 (0.15) | 0.32 (0.14)
  Negative Defocus Curve, -1.0 Diopter | 0.21 (0.14) | 0.17 (0.12)
  Negative Defocus Curve, -0.5 Diopter | 0.06 (0.11) | 0.02 (0.10)
  Negative Defocus Curve, 0.0 Diopter | -0.08 (0.07) | -0.10 (0.08)
  Positive Defocus Curve, 2.0 Diopter | 0.61 (0.11) | 0.57 (0.13)
  Positive Defocus Curve, 1.5 Diopter | 0.45 (0.13) | 0.44 (0.12)
  Positive Defocus Curve, 1.0 Diopter | 0.26 (0.13) | 0.27 (0.12)
  Positive Defocus Curve, 0.5 Diopter | 0.03 (0.11) | 0.02 (0.13)
  Positive Defocus Curve, 0.0 Diopter | -0.08 (0.08) | -0.09 (0.08)

ADVERSE EVENTS:
Description: There were no adverse events to report.
Arm/Group | ReSTOR Aspheric +4 | Acri LISA IOL
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/22
Other Adverse Events (participants affected / at risk) | 0/20 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No paper that incorporates Sponsor Condfidential information will be submitted for publication without Sponsor's prior written agreement.